CLINICAL TRIAL: NCT00974532
Title: Analysis of Calcium Balance in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 07-0959; G195
Record Dates: First submitted 2009-06-03; First posted 2009-09-10 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2009-09

CONDITIONS: Chronic Kidney Disease
Keywords: balance; chronic kidney disease; calcium; phosphorus
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Subjects with normal kidney function (Active Comparator): eGFR > 60 ml/min/m²
  Interventions: Dietary Supplement: High calcium diet 2000 mg/day; Dietary Supplement: Low calcium diet, 800 mg/day
- CKD late Stage 3 and Stage 4 (Experimental): eGFR 15-40 ml/min/m²
  Interventions: Dietary Supplement: High calcium diet 2000 mg/day; Dietary Supplement: Low calcium diet, 800 mg/day

INTERVENTIONS:
Dietary Supplement: High calcium diet 2000 mg/day — High calcium (2000 mg elemental calcium) diet x 9 days
Dietary Supplement: Low calcium diet, 800 mg/day — Low calcium (800 mg elemental calcium) diet x 9 days

SUMMARY:
Subjects with normal kidney function are able to excrete in their urine the calcium and phosphorus absorbed via the gastrointestinal tract and are thereby are able to maintain calcium and phosphorus balance. Patients with chronic kidney disease often have normal blood levels of calcium and phosphorus but no research has been conducted to determine if they are able to excrete their daily intake of these minerals. If they are not able to excrete their daily intake, these minerals could be deposited in soft tissue and blood vessels and contribute to the increased risk of cardiovascular disease seen in patients with chronic kidney disease. This study will determine if subjects with chronic kidney disease are in balance primarily with regard to calcium and at what level of kidney function they are no longer able to maintain balance. Understanding whether patients with chronic kidney disease are in balance will help direct future therapeutic interventions.

DETAILED DESCRIPTION:
We hypothesize that by Chronic Kidney Disease (CKD) late Stage 3 and Stage 4 patients are no longer able to maintain calcium balance by excreting their daily intake of calcium. We also hypothesize that the retention of calcium is not reflected in the serum concentration, as the body attempts to maintain the serum calcium concentration within narrow limits.

We will evaluate balance at two different levels of calcium intake. The two different levels were chosen to be at the extremes of normal calcium intake to provide insight into balance at low normal and high normal loads.

Specific expected experimental finding:

Directional Hypotheses:

Primary Hypothesis:

Late Stage 3/Stage 4 CKD patients (Estimated glomerular filtration rate [eGFR] 15-40 ml/min/m2) will excrete 20% of the absorbed calcium on the high calcium (2000 mg) diet. On the low calcium (800 mg) diet, CKD stage 4 patients will excrete 50% of the absorbed calcium. Gastrointestinal absorption will be 20% on both diets resulting in a net positive calcium balance of 320 mg on the high calcium intake and 80 mg on the lower calcium intake.

Subjects with normal kidney function (eGRF > 60 ml/min/m2) will excrete > 90% of the absorbed calcium on the high calcium diet and > 90% of the absorbed calcium on the low calcium diet. Gastrointestinal absorption will be 20% on both diets resulting in no net positive calcium balance on the high calcium intake or the lower calcium intake.

Secondary Hypothesis:

Late Stage 3/Stage 4 CKD patients (eGFR 15-40 ml/min/m2) will excrete 60% of their absorbed phosphorus on the 1600 mg phosphate diet. Normal subjects(eGRF > 60 ml/min/m2) will be expected to excrete > 90% of the absorbed phosphorus on the 1600 mg phosphate diet. Gastrointestinal phosphate absorption is expected to be 60% on both diets resulting in a net positive phosphorus balance of 192 mg and 384 mg in late stage 3/stage 4 CKD respectively. In addition, we hypothesize a decrease in fractional excretion of absorbed phosphorus as eGFR decreases.

The goal will be to study the following groups of patients:

1. Late Stage 3/Stage 4 CKD (eGFR 15-40 ml/min/m²)
2. Normal subject(eGFR > 60 ml/min/m²)

Estimated glomerular filtration rate (eGFR) will be calculated by the four variable Modification of Diet in Renal Disease (MDRD) equation which includes the serum creatinine, patients' age, gender and ethnicity.

Subjects with CKD will be recruited from the clinical practices of the nephrology division at the University of Colorado Health Sciences Center (HSC) by their nephrologists who will screen them for stable CKD based on historical laboratory data.

Following informed consent and prior to the start of the study, patients will be evaluated to determine whether they are vitamin D replete. Vitamin D deficiency is common not only in the elderly and chronically ill, but also in young healthy adults, especially at the end of winter. In a study of young healthy adults, ages 18 to 29, 36% of 69 subjects were found to be dihydroxy-vitamin D (Vitamin D 25-OH) deficient at the end of winter compared with 4% by the end of summer (13). For this reason, all patients will be assessed for Vitamin D 25-OH repletion prior to initiating the study diets.

This will be accomplished by checking serum Vitamin D 25-OH levels in all patients. Those with Vitamin D 25-OH levels less than 30 ng/mL will receive ergocalciferol 50,000 IU per week x 4 week. This is the Kidney Disease Outcome Quality Initiative (KDOQI) guideline recommendation for patients with CKD who are vitamin deficient. After that time, their Vitamin D 25-OH levels will be checked again to assess whether they are replete (i.e., serum level > 30 ng/mL). If their serum level is again below 30 ng/mL, a second 4 week course of ergocalciferol will be given. If the patient's serum Vitamin D 25-OH level remains < 30 ng/mL they will be excluded from further study. Once replete, subjects will remain on 50,000 IU ergocalciferol monthly throughout the study. This will ensure that vitamin D substrate is not a limiting factor in these patients. In addition the following medications will be discontinued following informed consent and for at least 1 month prior to the start of the first controlled diet, and for the duration of the study: paricalcitol, doxercalciferol, rocaltrol, cinacalcet, calcium supplements including calcium containing vitamins, or phosphate binders. Once patients are vitamin D replete they will have their calcium and phosphorus determined and be excluded from the study if their phosphorus exceeds 4.5 mg/dL or their calcium is outside the normal range.

Patients will be placed on two diets in random order for 9 days each. Randomization to diets will be accomplished using Permuted blocks stratified by CKD stage. Patients will receive one of two diets for each 9 day period, and then will subsequently go on the second diet after at least a one week "washout period". This wash-out period may last up to 4 weeks to accommodate a patient's schedule or to study menstruating women during the same phase of their cycle. Both patients and researchers will be blinded as to which diet the patients are receiving.

The last two days of each study period, patients will be admitted to the GCRC where they will collect two consecutive 24 hour urines for calcium, phosphorus, sodium, and creatinine, as well as a stool sample (see below) for calcium and phosphorus. The stool analysis for calcium and phosphorus will be used to determine the amount of the ingested calcium and phosphorus that is absorbed from the diet (fractional absorption), while the urinary calcium and phosphorus will be used to determine the fraction of absorbed mineral excreted in the urine. The urine sodium will be used to ensure stable dietary intake while the urinary creatinine will be used to ensure that the urine collections are complete and to determine the tubular reabsorption of phosphorus. A non-absorbable stool marker (Brilliant Blue) will be administered to patients on the evening of their admission to the GCRC and again the second evening in order to demarcate the time period over which the stool collected was formed. If the patient has not passed the second marker by the end of the 48 hour period, they will be asked to collect their stools at home and then bring them back to the General Clinical Research Center (GCRC).

On the final day of the patients' GCRC admission, after collection of the second 24 hour urine sample is complete, a final small urine collection will be obtained. This last urine sample will be used to measure spot calcium and phosphorus concentrations in order to compare these values to the known amount excreted in the two previous 24 hour collections.

Patients will also have a small saliva sample, approximately 3 mL, collected during their GCRC admission that will be used to measure salivary phosphorus concentration. These saliva samples will be stored at the GCRC until a laboratory has been identified to perform this testing.

Patients will also have an overnight fasting serum calcium, phosphorus, creatinine, 1,25 vitamin D, 25 vitamin D, intact Parathyroid hormone (PTH), and fibroblast growth factor (FGF) 23 levels measured at the completion of each 24 hour urine collection. In addition, patients will have a serum phosphorus determination prior to their evening meal on both evenings of their GCRC stay. After a "wash-out" period of at least one week patients will start the second week-long diet, at the end of which they will be admitted to the GCRC for a two day period. Patients may schedule their second diet period and GCRC stay within one to four weeks of the previous diet and GCRC stay at their convenience. The diets will be prepared by the GCRC nutrition staff.

Diet #1 (high-calcium diet):

Elemental calcium 2000 mg, phosphorus 1600 mg

Diet#2 (low-calcium diet):

Elemental calcium 800 mg, phosphorus 1600 mg

The diets will have the same sodium and potassium concentrations, and will be diabetic 2000 kilocalorie (kCal)/ day diets. As the goal of this study is to focus on calcium balance, which should not be affected by energy balance, there will be no adjustment for individuals who are in negative or positive energy balance. During their stay in the GCRC subjects will drink only deionized water or other beverages whose calcium and phosphorus content has been included in the assessment of dietary calcium intake.

All study subjects will be counseled to only eat food prepared for the study protocol. They will also be counseled to attempt to eat all of the food provided. They will be instructed to bring in any food that is not consumed. They will also be asked to keep a diet history of any food they eat that is not on the prepared diet. No supplemental vitamins, calcium, vitamin D, or phosphate binders will be taken during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age or greater and able to comply with the study protocol.
* eGFR within appropriate target ranges (15-40 ml/min/m² for late stage CKD stage 3 stage 4, and eGFR > 60 ml/min/m² for normal subjects)
* Stable kidney function defined as an eGFR which remains within a 10ml/min range over a 3 to 6 month period prior to study enrollment. This will be determined from historical laboratory data.
* Willing to follow study protocol
* Have a level of understanding and willingness to cooperate with all visits and procedures as described by the study personnel
* Overall stable medical condition, defined as no malignancy, metabolic condition or gastrointestinal condition that would make it difficult to comply with the study protocol and complete both dietary study periods
* Able to read the consent form and provide informed consent.
* Serum calcium and phosphorus within the normal range off of vitamin D analogues, calcium supplements, and phosphate binders for 1 month.

Exclusion Criteria:

* 1. Age less than 18 years
* Are pregnant, plan on becoming pregnant during the study period, or breast-feeding, if female.
* Patient declines participation.
* GI malabsorption, short bowel syndrome, frequent vomiting, or gastroparesis.
* Subject receiving synthetic parathyroid hormone, glucocorticoids, calcitonin or bisphosphonates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Calcium balance | 48 hour

SECONDARY OUTCOMES:
Phosphorus balance | 48 hours
PTH | 2 WEEKS
FGF-23 | 2 WEEKS

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Denver Health Sciences Center, Denver, Colorado, United States

REFERENCES:
- [Result] Spiegel DM, Brady K. Calcium balance in normal individuals and in patients with chronic kidney disease on low- and high-calcium diets. Kidney Int. 2012 Jun;81(11):1116-22. doi: 10.1038/ki.2011.490. Epub 2012 Feb 1. PMID 22297674